CLINICAL TRIAL: NCT05109663
Title: A Single-Centre, Single-Administration, Dose-Escalation Study and A Single-Centre, Randomized, Open-Label, Two-cycle Crossover Food Effect Study of SKLB1028 in Healthy Subjects
Brief Title: A Dose Escalation and Food Effect Study of SKLB1028 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HA114-CSP-006
Record Dates: First submitted 2021-10-27; First posted 2021-11-05 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-01

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — SKLB1028

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose Escalation Cohort 1: single oral dose of SKLB1028 (Experimental): Eligible subjects received a single dose of SKLB1028 50 mg on Day 1.
  Interventions: Drug: SKLB1028
- Dose Escalation Cohort 2: single oral dose of SKLB1028 (Experimental): Eligible subjects received a single dose of SKLB1028 100 mg on Day 1.
  Interventions: Drug: SKLB1028
- Food Effect Cohort A: SKLB1028, fasted dosing followed by fed dosing (Experimental): Eligible subjects received a single dose of SKLB1028 150 mg on Day 1 in a fasting state, and a single dose of SKLB1028 150 mg on Day 11 in a fed state, with a 10-day washout period between the 2 doses.
  Interventions: Drug: SKLB1028
- Food Effect Cohort B: SKLB1028, fed dosing followed by fasted dosing (Experimental): Eligible subjects received a single dose of SKLB1028 150 mg on Day 4 in a fed state, and a single dose of SKLB1028 150 mg on Day 14 in a fasting state, with a 10-day washout period between the 2 doses.
  Interventions: Drug: SKLB1028

INTERVENTIONS:
Drug: SKLB1028 — SKLB1028, capsule, oral

SUMMARY:
The purpose of this study was to explore the safety, tolerability and pharmacokinetics (PK) of single ascending oral doses of SKLB1028 in healthy subjects. This study has also explored the effect of food on the PK of SKLB1028.

DETAILED DESCRIPTION:
The study was divided into 2 parts. Part 1(Dose Escalation) included 2 cohorts (Cohort 1 and Cohort 2) and subjects received a single oral dose of SKLB1028 50 or 100 mg on Day 1. In Part 2 (Food Effect) included 2 cohorts (Cohort A and Cohort B), subjects received a single oral dose of SKLB1028 150 mg in a fasting and a fed state, with a 10-day washout period between the 2 doses.

ELIGIBILITY:
Inclusion Criteria:

-

Healthy subjects:

1. Male or female subjects aged 18 to 45 (including 18 and 45 years old), and the proportion of single sex should not be less than 1/3;
2. Male weight ≥50.0 kg, female weight ≥45.0 kg; body mass index (BMI) 18-24 kg/m^2 (inclusive);
3. Normal or abnormal results without clinically significance on all tests including medical history, physical examination, vital signs, clinical laboratory tests (routine blood test, blood biochemistry, routine urine test, coagulation function), etc;
4. Subjects are willing to use effective non-hormonal contraceptives such as condom and intrauterine device without medication, and not allowed to donate sperm from screening to the 6 months after the last dose administration unless permanent contraception has been taken, such as bilateral tubal ligation and vasectomy;
5. Voluntarily sign the informed consent form, and be willing to comply with the protocol.

Exclusion Criteria:

1. Previous or current clear psychiatric/neurological systems diseases; previous or current severe diseases, such as cardiovascular, liver and kidney, endocrine, respiratory, hematological, digestive and immune systems diseases; previous or current malignant tumors;
2. Allergic constitution, including a history of allergy to one or more medications, or other known severe allergic reactions;
3. Inability to swallow oral medications; previous or current diseases that may affect the absorption, distribution, metabolism, or excretion of the drug, or affect the evaluation of efficacy and safety of the drug, such as active bowel disease, partial or complete bowel obstruction and chronic diarrhea;
4. Previous or current diseases such as gastrointestinal ulcer and related bleeding;
5. Abnormalities of clinical significance in electrocardiogram (such as QTcF≥450 ms in males or ≥470 ms in females) or history of prolonged QTcF interval;
6. Any abnormalities of clinical significance in vital signs;
7. Any positive test result of hepatitis B surface antigen or hepatitis C virus antibody, or anti-human immunodeficiency virus antibody or anti-Treponema pallidum specific antibody;
8. Use of any prescription drugs, over-the-counter drugs, biologicals, proprietary Chinese medicine, herbal medicine, dietary supplements, health products, long-acting oral contraceptives or implantable long-acting contraceptives within 2 weeks prior to screening;
9. Use of any strong inhibitors or inducers of CYP3A4, CYP2C8 or P-gp within 2 weeks prior to screening;
10. Average daily intake of alcohol more than 14 units (14 units ≈285 mL of beer, or 25 mL of liquor, or 150 mL of wine) within 4 weeks prior to signature of informed consent, or a positive ethanol breath test at screening;
11. Smoking more than 5 cigarettes per day within 6 months prior to screening;
12. History of drug abuse within 1 year prior to screening, or positive urine drug screen at screening;
13. Average daily consumption of too much caffeinated beverages and foods or that might affect drug metabolism, such as coffee (over 1100 mL per day), tea (over 2200 mL per day), cola (over 2200 mL per day), functional beverage (over 1100 mL per day), chocolate (over 510 g per day) within 4 weeks prior to screening;
14. Consumption of cigarettes, alcohol or methylxanthine-rich food or beverage (such as coffee, tea, cola, chocolate, energy drinks) within 48 h before the administration, or those who have special dietary requirements and cannot follow a uniform diet;
15. Difficulty in venous blood collection or subjects with a history of fainting needle or blood;
16. Blood donation (or blood loss) ≥200 mL within 4 weeks prior to the screening, or who have a blood donation plan during the entire study or within 1 months after the study;
17. Subjects who have previously undergone surgery within 6 months prior to screening or who have a scheduled surgical plan (including cosmetic surgery, dental surgery and oral surgery) during the study period;
18. Participation in another clinical trial within 3 months before screening (whichever is administrated);
19. Any condition that the investigator considers inappropriate for participation in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events (TEAEs) | Throughout the study period, with an average of 10 days.
  TEAEs were assessed by CTCAE v5.0 in Part 1
Maximum plasma concentration (Cmax) of SKLB1028 in Part 2 | Pre-dose and multiple timepoints up to 144 hours post-dose
Area under the concentration-time curve from time 0 to last quantifiable concentration (AUC0-last) of SKLB1028 in Part 2 | Pre-dose and multiple timepoints up to 144 hours post-dose
Area under the concentration-time curve from time 0 to infinity (AUCinf) of SKLB1028 in Part 2 | Pre-dose and multiple timepoints up to 144 hours post-dose
Time to Cmax (Tmax) of SKLB1028 in Part 2 | Pre-dose and multiple timepoints up to 144 hours post-dose
Terminal-elimination half-life (T1/2) of SKLB1028 in Part 2 | Pre-dose and multiple timepoints up to 144 hours post-dose
Apparent volume of distribution (Vz/F) of SKLB1028 in Part 2 | Pre-dose and multiple timepoints up to 144 hours post-dose
Apparent clearance (CLz/F) of SKLB1028 in Part 2 | Pre-dose and multiple timepoints up to 144 hours post-dose

SECONDARY OUTCOMES:
Maximum plasma concentration ( Cmax) of SKLB1028 in Part 1 | Pre-dose and multiple timepoints up to 144 hours post-dose
Area under the concentration-time curve from time 0 to last quantifiable concentration (AUC0-last) of SKLB1028 in Part 1 | Pre-dose and multiple timepoints up to 144 hours post-dose
Area under the concentration-time curve from time 0 to infinity (AUCinf) of SKLB1028 in Part 1 | Pre-dose and multiple timepoints up to 144 hours post-dose
Time to Cmax (Tmax) of SKLB1028 in Part 1 | Pre-dose and multiple timepoints up to 144 hours post-dose
Terminal-elimination half-life (T1/2) of SKLB1028 in Part 1 | Pre-dose and multiple timepoints up to 144 hours post-dose
Apparent volume of distribution (Vz/F) of SKLB1028 in Part 1 | Pre-dose and multiple timepoints up to 144 hours post-dose
Apparent Clearance (CLz/F) of SKLB1028 in Part 1 | Pre-dose and multiple timepoints up to 144 hours post-dose
Number of participants with TEAEs | Throughout the study period, with an average of 20 days
  TEAEs were assessed by CTCAE v5.0 in Part 2

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, China